CLINICAL TRIAL: NCT02214576
Title: Observational Study of High Flow Nasal Canula Oxygen to Preoxygenate ARDS Patients That Require Intubation
Brief Title: High Flow Nasal Canula Oxygen Helps Preoxygenate ARDS Patients
Acronym: HIGHER
Status: Completed | Type: Observational
Sponsor: Hôpital Louis Mourier (Other)
Responsible Party: Principal Investigator, Prof Jean-Damien RICARD, Professor of Intensive Care Medicine, Assistant-head of ICU, Hôpital Louis Mourier
Other Study IDs: HLM_JDR2
Record Dates: First submitted 2014-08-11; First posted 2014-08-12 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Respiratory Distress Syndrome, Adult; intubation, intratracheal; Oxygen Inhalation Therapy; Positive-Pressure Respiration; laryngoscopy
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Tracheal intubation in the ICU is associated with significant complications and morbidity. Desaturation is among the most frequent and hazardous complication, occurring in almost one out of four intubations, that may in some instances lead to cardiac arrest; despite appropriate preoxygenation. Non-invasive ventilation may help improve preoxygenation but does not allow for apneic oxygenation and may not be performed in patients with neurological impairment. High flow nasal canula oxygen is increasingly used in the ICU in patients with acute hypoxemic respiratory failure and may be used to improve preoxygenation. It is currently used in our ICU for that purpose. Because high flow nasal canula oxygen is our first line oxyten therapy for patients with acute respirtory distress syndrome, we sought to determine its use as a means to ensure preoxygenation in those ARDS patients that require intubation.

DETAILED DESCRIPTION:
High flow nasal canula oxygen is increasingly used to provide heated and humidified oxygen in patients with acute respiratory failure. One of the major advantages of high flow nasal canula oxygen is the possibility to maintain oxygenation during laryngoscopy and thereby providing high flow apneic oxygenation. In addition, and contrary no non-invasive ventilation, preoxygenation may be used in patients with neurological impairment. Finally, the interest of this device is that it is the same that is maintained throughout the whole management of the patient, from ICU admission to intubation.

ELIGIBILITY:
Inclusion Criteria:

* ARDS according to the Berlin criteria
* use of high flow nasal canula oxygen

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute respiratory distress syndrome patients that require tracheal intubation in the ICU
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | 30 minutes
  oxygen saturation measured by pulse oxymetry during intubation and compared to levels before intubation

SECONDARY OUTCOMES:
complications | 60 minutes
  arrhythmia, hypotension, profound desaturation, cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien RICARD, MD, PhD, Principal Investigator — University Paris Diderot and Assistance Publique - Hôpitaux de Paris
Locations (1):
- Medico-surgical ICU, Louis Mourier Hospital, Colombes, France

REFERENCES:
- [Background] Ricard JD. High flow nasal oxygen in acute respiratory failure. Minerva Anestesiol. 2012 Jul;78(7):836-41. Epub 2012 Apr 24. PMID 22531566
- [Background] Sztrymf B, Messika J, Bertrand F, Hurel D, Leon R, Dreyfuss D, Ricard JD. Beneficial effects of humidified high flow nasal oxygen in critical care patients: a prospective pilot study. Intensive Care Med. 2011 Nov;37(11):1780-6. doi: 10.1007/s00134-011-2354-6. Epub 2011 Sep 27. PMID 21946925
- [Background] Sztrymf B, Messika J, Mayot T, Lenglet H, Dreyfuss D, Ricard JD. Impact of high-flow nasal cannula oxygen therapy on intensive care unit patients with acute respiratory failure: a prospective observational study. J Crit Care. 2012 Jun;27(3):324.e9-13. doi: 10.1016/j.jcrc.2011.07.075. Epub 2011 Sep 29. PMID 21958974
- [Background] Messika J, Ben Ahmed K, Gaudry S, Miguel-Montanes R, Rafat C, Sztrymf B, Dreyfuss D, Ricard JD. Use of High-Flow Nasal Cannula Oxygen Therapy in Subjects With ARDS: A 1-Year Observational Study. Respir Care. 2015 Feb;60(2):162-9. doi: 10.4187/respcare.03423. Epub 2014 Nov 4. PMID 25371400